CLINICAL TRIAL: NCT03036787
Title: Is There Any Differences in Motor And Cognitive Development Between Preterm (<37 Weeks) and Early Preterm (<32 Weeks) Infants? Two Years Follow Up Study
Brief Title: Is There Any Differences in Motor and Cognitive Development Between Preterm and Early Preterm Infants?
Status: Withdrawn | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Research Assistant, Gazi University
Other Study IDs: 11223
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Premature Baby
Keywords: Premature Baby; motor development; cognitive development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- moderate-early preterm infants: infant who births in 32 weeks to 37 weeks with family based intervention
  Interventions: Behavioral: family based intervention
- extremely-very preterm infants: infant who births in 27 weeks to 32 weeks with family based intervention
  Interventions: Behavioral: family based intervention

INTERVENTIONS:
Behavioral: family based intervention — behavioural advises to family for normal motor development

SUMMARY:
Infant born preterm have an increased risk of adverse long-term developmental outcomes.The risk associated with preterm birth increase as gestational age decreases, and vulnerability remains in extremely- very preterm (<32 weeks) and moderate- late preterm (>32 weeks). There are many studies in the literature showed that the prevalence of developmental delay increases with premature birth. However, there is no study in the literature investigates long term follow up motor and cognitive development in subgroups of preterm infants . Hence the aim of this study is to evaluate the differences in motor and cognitive development in moderate-late (>32 weeks) and extremely-very preterm infants.

DETAILED DESCRIPTION:
A convenience of infants with premature birth recruiting from Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation. Babies divide into two groups according to the gestational ages. Babies with gestational ages between 32-36 weeks and 6 days (including the given days) are categorized as moderate-late preterm, while those born before 32 weeks are grouped as extremely and very preterm. Each group contains 20 babies. First, sociodemographic information and histories of babies are obtaining. Ages and contact information of the parents are recording. Prenatal and natal risk factors of the mothers are querying. Gestational ages and height, weight, and head circumferences of babies at birth are recording. Number of pregnancies, live births and abortions, type of delivery, multiple pregnancies for mothers as well as consanguinity between parents are asking.The Alberta Infant Motor Scale is using to evaluate spontaneous motor movements of the baby. It evaluates the baby at prone, supine, sitting, and standing positions. Bayley Scales of Infant and Toddler Development scales screen for cognitive, language, and motor development in babies. All infants will be testing in 3-6-9-12-15-18-24 months of ages.

ELIGIBILITY:
Inclusion Criteria:

* adjusted age of 24 months or less, born with a gestational age of 36 weeks and 6 days or earlier, not having any systemic disease, and accepting to join the study

Exclusion Criteria:

* age greater than 24 months and born with a gestational age of 37 weeks or more
* having major risk factor

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm infants born with <37 weeks.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-02-09 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Motor development assessed with the Alberta Infant Motor Scale | Each 3 months from beginning to two years
  The Alberta Infant Motor Scale is going to use

SECONDARY OUTCOMES:
Cognitive development assessed with the Bayley Scales of Infant and Toddler Development | Each 3 months from beginning to two years
  Bayley Scales of Infant and Toddler Development

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Phd, Study Chair — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We have no decided yet